CLINICAL TRIAL: NCT00817336
Title: Effect of an NMDA-based Intervention on Biomarker Measures of Cognitive Dysfunction in Schizophrenia
Brief Title: Biomarkers in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08I/C19-0
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: biomarker; EEG; schizophrenia; NMDA; D-serine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-serine (Experimental): 60 mg/kg/day
  Interventions: Drug: D Serine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D Serine — 60 mg/kg/day
  Arms: D-serine
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
N-methyl-D-aspartate (NMDA)-type glutamate receptors are thought to play a pivotal role in neurocognitive dysfunction associated with schizophrenia. Further, several novel glutamate-based classes of compound are presently in development as potential novel treatments for persistent negative and cognitive symptoms. The study will assess effectiveness of a NMDA-based intervention on biomarkers related to schizophrenia as a mechanism for developing appropriate outcome batteries for future trials of novel compounds.

DETAILED DESCRIPTION:
16 in- or outpatients with DSM-IV-TR schizophrenia or schizoaffective disorder and prominent negative symptoms will be recruited for this study. This study will consist of a randomized trial of D-serine (60 mg/kg/d) vs. placebo using a crossover design with a 2-week baseline lead-in, and two 6-week intervention arms separated by a two week, placebo controlled washout period. Biomarkers will be assessed at baseline for each treatment arm, acutely (day 7) following treatment initiation, and following 6 weeks of treatment (6 biomarker sessions total). Primary biomarker outcome measures will include 1) amplitude of the mismatch negativity (MMN) waveform and 2) amplitude of the visual P1 potential. Symptomatic outcome measures will include PANSS and composite score of the MATRICS neuropsychological battery. The study will be supported from ongoing NIMH-funded Cooperative Drug Development Grant (CDDG) to the PI.

ELIGIBILITY:
Inclusion criteria:

* Age 18-64
* SCID diagnosis of Schizophrenia or Schizoaffective Disorder.
* PANSS 3 factor negative symptom (screening and baseline visit 1 and visit 3) score of >20 and PANSS total score between 60-110. Any degree of positive symptoms is acceptable but the total PANSS score must not exceed 110.
* SAS total score less than or equal to 12 and a Calgary Depression Inventory total score less than or equal to 10 and suicide (item 8) less than moderate (<2).
* Two consecutive CGI ratings at screening and baseline (visit 1 and 3) with no change in score.
* Estimated Glomerular Filtration Rate (GFR)(a measure of renal function) greater than or equal to 60.

Exclusion criteria:

* Organic brain disorder, including epilepsy; mental retardation; or a medical condition whose pathology or treatment would likely alter the presentation or treatment of schizophrenia or significantly increase the risk associated with any of the proposed treatments
* Current DSM-IV diagnosis of drug/alcohol abuse in last month and current DSM-IV diagnosis of drug/alcohol dependence in last 6 months
* Pregnant female patients
* Impaired renal function
* Significant extrapyramidal symptoms (as reflected by a total score of 10 or above on the SAS scale), and depressive symptoms (as reflected by a score of 10 or above on the Calgary Depression Scale for Schizophrenia)
* Patients who are unable to or unwilling to participate in the Cognitive assessment (MATRICS) and the electrophysiology tasks .
* Patients on clozapine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Javitt, MD, PhD, Principal Investigator — New York University
Locations (1):
- Nathan Kline Institute, Orangeburg, New York, United States

REFERENCES:
- [Derived] Kantrowitz JT, Epstein ML, Lee M, Lehrfeld N, Nolan KA, Shope C, Petkova E, Silipo G, Javitt DC. Improvement in mismatch negativity generation during d-serine treatment in schizophrenia: Correlation with symptoms. Schizophr Res. 2018 Jan;191:70-79. doi: 10.1016/j.schres.2017.02.027. Epub 2017 Mar 18. PMID 28318835

RESULTS

PARTICIPANT FLOW:
Groups:
- D-serine Followed by Placebo; Placebo Followed by D-serine: subjects received a fixed dose of D-serine 60 mg/kg/day in a randomized, placebo-controlled crossover study of d-serine and placebo each for 6 weeks. Subjects were randomly assigned to receive (d-serine or placebo) in the first treatment phase, followed by two-weeks of single-blind placebo, which was followed by the alternative treatment in a second-phase.
Period: Overall Study
Arm/Group | D-serine Followed by Placebo | Placebo Followed by D-serine
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: There were no statistically significant differences by treatment order
Groups:
- D-serine Followed by Placebo; Placebo Followed by D-serine: Does not include 1 drop-out during phase 1
- Total: Total of all reporting groups
Arm/Group | D-serine Followed by Placebo | Placebo Followed by D-serine | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 44.6 (11) | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 7 | 13
In-patient number [Count of Participants; unit: Participants] | 6 | 4 | 10
Chlorpromazine equivalents [Mean (Standard Deviation); unit: mg] | 1135 (967) | 795 (496) | 965 (760)
PANSS total [Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Symptom Scale (PANSS) range from 30-210, with higher scores worse
  units on a scale | 83.7 (9) | 80.1 (10) | 80.8 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: PANSS Total
Description: Positive and Negative Symptom Scale (PANSS) range 30-210
Time Frame: 6 weeks
Population: Final score end of six weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale | 77.9 (9.3) | 80 (10.3)
Statistical Analysis 1: Comparison: D-serine vs Placebo; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Cohen's d = 0.80

2. Primary Outcome: MMN Amplitude
Description: Final MMN amplitude
Time Frame: 6 weeks
Population: Includes 11 subjects with analyzable MMN data
Measure: Mean (Standard Deviation); unit: micro volts
Arm/Group | D-serine | Placebo
Number analyzed (Participants) | 11 | 11
micro volts | -1.21 (.6) | -.21 (.9)
Statistical Analysis 1: Comparison: D-serine vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Cohen's d = 2.3

3. Secondary Outcome: MATRICS
Description: MATRICS assessing 7 domains (Speed of Processing, Attention/Vigilance, Working Memory, Verbal Learning, Visual Learning, Reasoning and Problem Solving, and Social Cognition. Raw scores are converted into a composite T-score (normative mean = 50; standard deviation = 10), where higher values indicated less impairment.
Time Frame: 6 weeks
Population: Final score after six weeks
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | D-serine | Placebo
Number analyzed (Participants) | 14 | 14
T score | 26.2 (7.6) | 25.7 (7.9)
Statistical Analysis 1: Comparison: D-serine vs Placebo; Test type: Superiority or Other; p = .31, Mixed Models Analysis; Cohen's d = 0.41

4. Secondary Outcome: Visual P1
Time Frame: 6 weeks
Population: includes subjecst with valid visual p1 data
Measure: Mean (Standard Deviation); unit: micro volts
Arm/Group | D-serine | Placebo
Number analyzed (Participants) | 12 | 12
micro volts | -.21 (1.3) | -.54 (1.2)
Statistical Analysis 1: Comparison: D-serine vs Placebo; Test type: Superiority; p = .41, Mixed Models Analysis; Cohen's d = 0.41

ADVERSE EVENTS:
Description: per intervention
Groups:
- D-serine/Placebo Crossover: subjects received a fixed dose of D-serine 60 mg/kg/day in a randomized, placebo-controlled crossover study of d-serine and placebo each for 6 weeks. Subjects were randomly assigned to receive (d-serine or placebo) in the first treatment phase, followed by two-weeks of single-blind placebo, which was followed by the alternative treatment in a second-phase.
Arm/Group | D-serine/Placebo Crossover
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes